CLINICAL TRIAL: NCT03194399
Title: Development of Personalized Health Care Service in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Eun Joo Yang, Study Chair, Seoul National University Bundang Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-1509-314-002
Record Dates: First submitted 2017-06-07; First posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer; Lymphedema; Cancer-related Problem/Condition
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breast cancer patients (Experimental)
  Interventions: Behavioral: Personalized health care service

INTERVENTIONS:
Behavioral: Personalized health care service — Physical activity coaching, other functional outcome observation

SUMMARY:
In order to develop effective personalized healthcare service program for breast cancer rehabilitation, we designed this study using mobile phone and clinical intervention(feedback coaching).

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patient (age over 18), Cancer stage under 3, Android OS smartphone user

Exclusion Criteria:

* Cancer stage over 4, Patients diagnosed with multiple cancer, Patient who can not participate rehabilitation exercise program

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-11-27 (Actual); Primary Completion 2016-02-15 (Actual); Study Completion 2016-02-22 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction change | Baseline and after 2 weeks, 4 weeks of lifestyle modification
  Patient subjective evaluation by survey on satisfaction

SECONDARY OUTCOMES:
Physical activity change | Baseline and after 2 weeks, 4 weeks of lifestyle modification
  Physical activity measurement by step count
Functional outcome change | Baseline and after 2 weeks, 4 weeks of lifestyle modification
  (Physical)Functional outcome measurement by breast cancer patient questionnaire
Quality of care change | Baseline and after 2 weeks, 4 weeks of lifestyle modification
  Quality of care measurement by breast cancer patient questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Eunjoo Yang, PhD, Study Chair — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No